CLINICAL TRIAL: NCT04425499
Title: A Gamified Network for Surgical Education During COVID-19: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Érica Patocskai, Assistant professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CERSES 20-068-D
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Advanced Suturing Skills; Surgical Education
Keywords: Running subcuticular sutures; Surgical education; Advanced suturing skills; Distant learning; Peer-learning; Network

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Placebo Comparator): On GEN (Gamified Educational Network), each student will view individually eight videos of an expert performing a running subcuticular suture correctly. The OSATS (Objective Structured Assessment of Technical Skills) Global Rating Scale (GRS) and Subcuticular Suture Checklist will be available beside each video and students will be required to fill them out for each video. For three days, students will have access to a distinct set of videos on GEN to learn running subcuticular sutures. Three days later, students will view the same eight videos of an expert performing a running subcuticular suture, however, the videos will be shuffled in a different order. The order of the videos will be the same for all students.
  Interventions: Other: Learning running subcuticular sutures on the Gamified Educational Network
- Self-learning (Experimental): Each student will view eight videos individually and complete the GRS and Subcuticular Suture Checklist for each video. Six videos will contain errors and two videos will not. The errors will be technical mistakes in the execution of a running subcuticular suture. For three days, students will have access to a distinct set of videos on GEN to learn running subcuticular sutures. Three days later, all students will repeat this activity. However, the same videos will be shuffled in a different order. The order of the videos will be the same for all students.
  Interventions: Other: Learning running subcuticular sutures on the Gamified Educational Network
- Peer-learning (Experimental): Each student will view eight videos and complete the GRS and Subcuticular Suture Checklist for each video. Six videos will contain errors and two videos will not. After this initial test, students will interact with other medical students in their group on the GEN platform anonymously for three days. We will display distinct videos on GEN. Comments will be allowed in an interactive way to encourage exchanges. Students will be required to participate in the discussion of at least two videos. Students will not be able to modify their answers on the initial test. On the third day, students in this group will perform a post-test individually with the same eight initial videos but shuffled. The order of the videos will be the same for all students.
  Interventions: Other: Learning running subcuticular sutures on the Gamified Educational Network
- Peer-learning with expert feedback (Experimental): Same as group 3, the only difference is that an expert will actively participate in the discussion by commenting on each video on GEN, enhancing students' educational experience. Although anonymous, students will be able to identify the expert as the name "expert" will be used. The expert will answer any question and comment on the discussion in order to guide the students.
  Interventions: Other: Learning running subcuticular sutures on the Gamified Educational Network

INTERVENTIONS:
Other: Learning running subcuticular sutures on the Gamified Educational Network — Each arm will have 15 participants who will learn how to perform running subcuticular sutures through videos on GEN.

SUMMARY:
Background: Traditionally, medical students learn surgical skills through the observation of a resident or a surgeon performing the technique. Due to inconsistent practice opportunities in the clinical setting, a disparity of skill levels among students has been observed. In addition, the poor availability of faculty professors is a limiting factor in teaching and adequately preparing medical students for clerkship years. With the ongoing COVID-19 pandemic, medical students do not have access to traditional suturing learning opportunities. Didactic courses are available on videoconferencing platforms, but they do not include technical training.

Objective: Our overarching goal is to evaluate the efficacy of web-based peer-learning for advanced suturing techniques (i.e., running subcuticular sutures). The investigators will use GEN (Gamified Educational Network), a newly developed online learning tool. The investigators will assess students' ability to identify and to perform the right technique. The investigators will also assess students' satisfaction with regards to GEN.

Methods: The investigators will conduct a prospective randomized controlled trial with blinding of expert examiners. First-year medical students in the Faculty of Medicine of Université de Montréal will be randomized to four groups: 1) control group, 2) self-learning, 3) peer-learning, and 4) peer-learning with expert feedback. Each arm will have 15 participants who will learn how to perform running subcuticular sutures through videos on GEN. For our primary outcome, students' ability to identify the right technique will be evaluated before and after the intervention on GEN. They will view eight videos and rate the surgical technique using the OSATS (Objective Structured Assessment of Technical Skills) Global Rating Scale (GRS) and the Subcuticular Suture Checklist as evaluation criteria. For our secondary outcomes, students will anonymously record themselves performing a running subcuticular suture and will be evaluated using the same scales. Then, a survey will be sent to analyze the overall performance of the platform.

Results: The study will be conducted in accordance with the Declaration of Helsinki and has been approved by our institutional review board (CERSES 20-068-D). No participants have been recruited yet.

Conclusions: Peer-learning through GEN has the potential to overcome significant limitations related to the pandemic and the lack of availability of faculty professors. Further, a decrease of the anxiety related to traditional suturing classes can be expected. The investigators aim to create an innovative and sustainable method of teaching surgical skills to improve the efficiency and the quality of surgical training in medical faculties. With the current world events of COVID-19, the necessity for such tools are imperative.

ELIGIBILITY:
Inclusion Criteria:

* Students must be enrolled in their first year of medical school at Université de Montréal.

Exclusion Criteria:

* Students who have returned after a leave such as a sabbatical year/sick leave/maternity leave.
* Students who have already obtained a medical degree in another country.
* Students who studied medicine in another country.
* Any student injured at the beginning of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Retention of the correct technique for running subcuticular sutures | three days
  The Global Rating Scale and Subcuticular Suture Checklist will be used to measure

SECONDARY OUTCOMES:
Technical ability to perform a subcuticular suture | half a day
  The Global Rating Scale and Subcuticular Suture Checklist will be used to assess students' skills
Satisfaction with the GEN platform | five minutes
  A survey will be sent to students

REFERENCES:
- [Derived] Guerard-Poirier N, Meloche-Dumas L, Beniey M, Torres A, Kapralos B, Dhane M, Mercier F, Younan R, Dubrowski A, Patocskai E. The exploration of remote simulation strategies for the acquisition of psychomotor skills in medicine: a pilot randomized controlled trial. Discov Educ. 2023;2(1):19. doi: 10.1007/s44217-023-00041-2. Epub 2023 Jul 17. PMID 37469757
- [Derived] Guerard-Poirier N, Beniey M, Meloche-Dumas L, Lebel-Guay F, Misheva B, Abbas M, Dhane M, Elraheb M, Dubrowski A, Patocskai E. An Educational Network for Surgical Education Supported by Gamification Elements: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Dec 14;9(12):e21273. doi: 10.2196/21273. PMID 33284780